CLINICAL TRIAL: NCT06592755
Title: Single-Incision Gasless Endoscopic Total Thyroidectomy Via Subclavian Approach Versus Open Surgery for Papillary Thyroid Carcinoma
Brief Title: Single-Incision Gasless Endoscopic Total Thyroidectomy Via Subclavian Approach Versus Open Surgery for PTC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1124-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- the Subclavian Approach group: The patients chose to undergo total thyroidectomy and central compartment neck dissection via the single-incision subclavian approach.
  Interventions: Procedure: single-incision, gasless endoscopic total thyroidectomy with central compartment neck dissection
- the conventional open surgery group: The patients chose to undergo total thyroidectomy and central compartment neck dissection via the conventional open surgery approach.
  Interventions: Procedure: conventional open surgery

INTERVENTIONS:
Procedure: single-incision, gasless endoscopic total thyroidectomy with central compartment neck dissection — The included patients chose to undergo single-incision, gasless endoscopic total thyroidectomy with central compartment neck dissection via the subclavian approach based on patients preference.
  Groups: the Subclavian Approach group
Procedure: conventional open surgery — These patients chose to undergo total thyroidectomy with central compartment neck dissection via conventional open surgery based on patients preference.
  Groups: the conventional open surgery group

SUMMARY:
Historically, performing a contralateral thyroid lobectomy and lymph node dissection via the subclavian approach was considered challenging. This study aimed to evaluate the safety and feasibility of single-incision gasless endoscopic total thyroidectomy and central compartment neck dissection via the subclavian approach (SCA) in comparison to conventional open surgery for the treatment of papillary thyroid carcinoma (PTC) retrospectively.

DETAILED DESCRIPTION:
Historically, performing a contralateral thyroid lobectomy and lymph node dissection via the subclavian approach was considered challenging. This study aimed to evaluate the safety and feasibility of single-incision gasless endoscopic total thyroidectomy and central compartment neck dissection via the subclavian approach (SCA) in comparison to conventional open surgery for the treatment of papillary thyroid carcinoma (PTC) retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* (1) thyroid neoplasm <3.0 cm;
* (2) well differentiated papillary thyroid carcinoma.

Exclusion Criteria:

* (1) extrathyroidal extensions estimated in ultrasonography scan;
* (2) enlarged lymph nodes in lateral neck compartment on palpation, or US scan;
* (3) suspected distant metastases;
* (4) previous history of neck radiation therapy and/or surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients, who were diagnosed with papillary thyroid carcinoma at our center, chose to undergo either single-incision, gasless endoscopic total thyroidectomy with central compartment neck dissection via the subclavian approach or conventional open surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
the disease-free survival | up to 24 months
  The disease-free survival refers to the probability of survival without any biologic, structural, or functional events.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China